CLINICAL TRIAL: NCT00562679
Title: Long Term Effects of Sleep Apnea in Patients With Coronary Artery Disease
Brief Title: Coronary Artery Disease and Sleep Apnea
Status: Completed | Type: Observational
Sponsor: Umeå University (Other)
Collaborators: Swedish Heart Lung Foundation (Other); Norrländska Hjärtfonden (Unknown); Jämtland County Council, Sweden (Other Government)
Other Study IDs: 93-032
Record Dates: First submitted 2007-11-21; First posted 2007-11-22 (Estimated); Last update posted 2008-07-02 (Estimated); Status verified 2008-06

CONDITIONS: Coronary Artery Disease
Keywords: Patients with coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 2 groups: The cohort is grouped according to one group with sleep apnea and one group without sleep apnea
  Interventions: Other: There is no intervention

INTERVENTIONS:
Other: There is no intervention

SUMMARY:
The purpose of this study is to determine the effect of sleep apnea on mortality, stroke and myocardial infarction among 408 patients with coronary artery disease referred for evaluation of coronary intervention who were examined with overnight cardio respiratory monitoring between March 1992 and June 1995.

ELIGIBILITY:
Inclusion Criteria:

* Men and women younger than 70 with disabling angina pectoris and coronary disease according to coronary angiography.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patiens with coronary artery disease beeing referred for evaluation of coronary intervention
Sampling Method: Probability Sample
Enrollment: 408 (Actual)
Dates: Start 1992-03; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Stroke, death, acute myocardial infarction | 10 years from date of inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Mooe, MD, PhD, Principal Investigator — Dept Medicine, Östersund Hospital, Östersund
Locations (1):
- Dept of Cardiology, Umeå, Sweden

REFERENCES:
- [Derived] Valham F, Mooe T, Rabben T, Stenlund H, Wiklund U, Franklin KA. Increased risk of stroke in patients with coronary artery disease and sleep apnea: a 10-year follow-up. Circulation. 2008 Aug 26;118(9):955-60. doi: 10.1161/CIRCULATIONAHA.108.783290. Epub 2008 Aug 12. PMID 18697817